CLINICAL TRIAL: NCT00469885
Title: Harm Reduction Treatment for Smokers With Cardiovascular Disease {Reduction of Smoking in Cardiovascular Disease Patients (ROSCAP)}
Brief Title: Reduction of Smoking in Cardiac Disease Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Anne Joseph, UMN
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P50DA13333-8; NIDA P50 DA13333; P50DA013333 (NIH)
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2008-06

CONDITIONS: Cardiovascular Disease; Tobacco Use Disorder
Keywords: Smoking cessation; cardiovascular disease; smoking reduction; nicotine replacement
MeSH Terms: conditions — Cardiovascular Diseases; Tobacco Use Disorder; Smoking Cessation; Smoking Reduction | interventions — Nicotine Replacement Therapy; Nicotine; Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): Usual care
  Interventions: Behavioral: Motivational counseling
- 2 (Other): Reduction
  Interventions: Drug: Nicotine replacement

INTERVENTIONS:
Drug: Nicotine replacement — For reduction
  Other Names: Nicoderm, Nicorrette
  Arms: 2
Behavioral: Motivational counseling — No drugs
  Other Names: Behavioral counseling
  Arms: 1

SUMMARY:
This study evaluates the effect of smoking reduction vs usual care (quitting advice only) for individuals with peripheral arterial disease who smoke.

DETAILED DESCRIPTION:
This study randomly assigns smokers who do not have a quit date set to either a smoking reduction grop or usual care group. The smoking reduction group receives behavioral counseling on smoking reduction and nicotine patch and/or gum to reduce the number of cigarettes smoked per day by at least 50%. The usual care group is given brief advice to quit smoking and referral to local cessation services. To be included in the study, participants must have peripheral arterial disease (defined as ankle Brachial Index equal to or less than 0.85 or history of prior revascularization) and they must be daily smokers (defined as at least 1 cigarette, cigar, or tobacco pipe daily). Participants complete questionnaires that measure mood, functional ability, smoking history, and motivation to quit smoking. Participants will be followed in this study for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* To be included in the study, participants must have peripheral arterial disease (defined as ankle Brachial Index equal to or less than 0.85 or history of prior revascularization) and they must be daily smokers (defined as at least 1 cigarette, cigar, or tobacco pipe daily).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2001-01; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Number of cigarettes per day | 6 months
ASCVD health changes | 6 months
Days of abstinence from cigarettes | 6 months
Number of quit attempts | 6 months

SECONDARY OUTCOMES:
Withdrawal symptoms | ongoing through 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Anne Joseph, MD, Principal Investigator — Veteran's Administration Hospital
Locations (2):
- United States (2):
  - Univeristy of Minnesota, Minneapolis, Minnesota
  - Univerisity of Minnesota, Minneapolis, Minnesota